CLINICAL TRIAL: NCT05598554
Title: The Effects of Chair-Based Yoga With Telerehabilitation on Function and Quality of Life in Elderly Individuals
Brief Title: The Effects of Telerehabilitation And Chair-based Yoga In The Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevval Kadriye Bakir (Other)
Responsible Party: Sponsor-Investigator, Sevval Kadriye Bakir, Investigator, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 019
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Telerehabilitation; Chair-based Yoga; Elderly People
Keywords: depression; quality of life; quality of sleep; pain; chair-based yoga; Telerehabilitation
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Pain | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): chair-based yoga program with tele-rehabilitation was applied to elderly people.
  Interventions: Other: Telerehabilitation
- Control Group (Active Comparator): 1 session of training was given on the effect of physical activity and exercise on function and quality of life.
  Interventions: Other: information

INTERVENTIONS:
Other: Telerehabilitation — Chair-based yoga with telerehabilitation was applied to the study group for 45 minutes a day, 2 days a week, for 6 weeks.
  Arms: Study Group
Other: information — A one-session training was provided on the effects of exercise on quality of life.
  Arms: Control Group

SUMMARY:
The aim of the study is to investigate the effects of chair-based yoga with rehabilitation on quality of life is affected in elderly people. Depending on the changes in the body as a result of aging, people's quality of life is affected. In order to increase or protect the quality of life in elderly people, telerehabilitation practices are emphasized. Telerehabilitation is a promising system for the elderly thanks to its advantages.

As a practice, chair-based yoga, a modified form of yoga, was preferred. Chair-based yoga makes yoga more doable and safe for older people. Chair-based yoga with telerehabilitation was performed with the participants. Pain level, sleep status, functional capacity, quality of life, mental health and depression were followed by evaluations at the beginning and end of the process.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and over,
* Having a Standardized Mini Mental Test Score of 24 and above,
* physically active (self-sustaining),

Exclusion Criteria:

* severe cardiopathy,
* uncontrolled hypertension,
* mental disorder,
* Presence of any health condition that may prevent functional autonomy test such as hearing and vision,
* have mental disorders and dementia,
* people with any unstable medical condition

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test (SFT) | 6 weeks
  It is another test protocol in which the physical fitness of elderly people is evaluated with a few test parameters. SFT Test Protocol; It consisted of 6 stations including chair sit-stand, weight lifting, chair sit-down, 2-minute stepping, 8-step up-go and back scratching tests.
Nottingham Health Profile (NHP) | 6 weeks
  It is a general patient-reported outcome measure intended to measure subjective health status. It is a questionnaire designed to measure a patient's views on his or her health status in various fields. It can be completed in 5 minutes. NHP consists of two parts.

SECONDARY OUTCOMES:
Charlson Comorbidity Index | 6 weeks
  Scaling that can be applied by quantifying comorbidities and examining their effects on prognosis in clinical trials, with the informant or by obtaining information from medical records. 19 disease states are evaluated.
Barthel Index for Activities of Daily Living | 6 weeks
  Scaling with the informant to assess the physical adequacy of geriatric subjects and their independence in basic activities of daily living. 10 activities of daily living are evaluated. The Bartel index (BI) is a widely used scale in functional disability.
Mini Mental State Assessment | 6 weeks
  Screening test in which cognitive functions are evaluated globally. With the standardized mini mental test, the patient is evaluated under 5 main headings.
Yesavage Geriatric Depression Scale | 6 weeks
  Scaling applied to evaluate geriatric cases in terms of depressive mood. General mood characteristics such as attentional state, decision-making process, and perspective on the future are questioned.
Tinetti Balance and Gait Test | 6 weeks
  It is a scaling applied in the presence of an observer in order to evaluate the walking and balance abilities of the person. It consists of 16 questions. TDYD evaluates balance ability and gait under 2 main headings.
Clinical Frailty Scale | 6 weeks
  It is a scaling that can be done with the case itself or the caregiver in order to evaluate the cases in terms of fragility with clinical findings. It consists of 9 questions.
Pittsburgh Sleep Quality | 6 weeks
  It is a scale that evaluates sleep quality with a total of 19 questions under 7 main headings. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points.
Mc Gill Pain Questionnaire | 6 weeks
  It consists of four parts. In the first part, the patient is asked to mark the location of the pain on the body chart. Part Two: In this part, there are 20 sets of words that examine pain in terms of sensory, perceptual and evaluation. The patient is told to choose the word set that fits his pain and to mark the word that fits his pain in the chosen set. In the third part, the relationship of pain with time takes place. There are word groups to determine the continuity of pain, its frequency, and factors that increase/reduce pain. In the fourth part, five word groups ranging from "mild" pain to "unbearable" pain to determine the severity of pain; In addition, six questions were included to determine the severity of pain that the patient can accept or experience without discomfort, which is also defined as "experienceable=target pain".

CONTACTS AND LOCATIONS:
Overall Officials: Şevval Bakır, Principal Investigator — sevval.bak19@gmail.com; Gül D Yelvar, Study Director — guldenizy@yahoo.com
Locations (1):
- Istinye University Topkapi Campus, Istanbul, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No